CLINICAL TRIAL: NCT05798559
Title: Investigation of the Effectiveness of Sleep Hygiene Education in Mothers With Preschool Children: A Randomized Controlled Study
Brief Title: Sleep Hygiene Education in Mothers With Preschool Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, Zeynep Çorakcı Yazıcıoğlu, Principal Investigator, Bezmialem Vakif University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CORAKCİ-003
Record Dates: First submitted 2023-03-23; First posted 2023-04-04 (Actual); Last update posted 2023-08-24 (Actual); Status verified 2023-08

CONDITIONS: Sleep; Habits; Neurodevelopmental Disorders
Keywords: Sleep Hygiene; Neurodevelopmental Disorders
MeSH Terms: conditions — Habits; Neurodevelopmental Disorders; Sleep Hygiene

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
  Mothers of children with neurodevelopmental disorders will be included in the study.
  Inclusion criteria for the study:
  * Having a child with a neurodevelopmental disorder
  * Be over 18 years old and literate
  * Having a child(s) of pre-school age (3-6 years old)
  * Communicating and collaborating
  Intervention and study group will be formed by simple randomization.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): * "Sleep Training" will be applied.
  * With the training, examples will be presented to mothers that they can apply in their daily lives.
  * 1 month will be followed
  Interventions: Behavioral: Sleep Training
- Control Group (No Intervention): No training will be provided
  note: "Sleep Training" will be given after the study is completed so that the control group is not victimized.

INTERVENTIONS:
Behavioral: Sleep Training — These are the trainings given by the researchers in order to regulate the sleep routine and environment. Content will be presented to improve sleep processes by arranging living habits.
  Arms: Intervention Group

SUMMARY:
The goal of this clinical trial is to gain importance of sleep routine and environment in mothers have children with neurodevelopmental disorders. The main questions it aims to answer are:

* What is the importance of sleep routine and environment in children with neurodevelopmental disorders?
* What kind of an effect does the awareness that mothers gain through sleep trainings have?

Participants will:

* Evaluations will be applied to all participants
* Divided into intervention and control groups
* The intervention group will be given "Sleep Training" and followed up for about 1 month.
* The results between the two groups will be compared

Researchers will compare intervention and control groups to see if turning a healthy sleep routine into a life habit

ELIGIBILITY:
Inclusion Criteria:

* Having a child with a neurodevelopmental disorder
* Be over 18 years old and literate
* Having a child(s) of pre-school age (3-6 years old)
* Communicating and collaborating

Exclusion Criteria:

* Having a neurological or psychiatric disease that prevents communication and cooperation

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — To be a mother
Enrollment: 35 (Actual)
Dates: Start 2023-06-05 (Actual); Primary Completion 2023-08-15 (Actual); Study Completion 2023-08-23 (Actual)

PRIMARY OUTCOMES:
The Children's Sleep Habits Questionnaire | 1 month
  Questionnaire that has been used in a number of studies to examine sleep behavior in young children. The Questionnaire includes items relating to a number of key sleep domains that encompass the major presenting clinical sleep complaints in this age group: bedtime behavior and sleep onset; sleep duration; anxiety around sleep; behavior occurring during sleep and night wakings; sleep-disordered breathing; parasomnias; and morning waking/daytime sleepiness.

SECONDARY OUTCOMES:
Occupational Balance Questionnaire | 1 month
  The purpose of the questionnaire is to measure satisfaction according to the amount and variety of daily activities of the individual and to define their occupational balance according to the obtained results.

CONTACTS AND LOCATIONS:
Overall Officials: Kardelen Yıldırım, Lecturer, Study Chair — Bezmialem Vakif University; Gülşah Zengin, Lecturer, Study Director — Bezmialem Vakif University; Sultan Akel, Lecturer, Study Director — Bezmialem Vakif University; Sümeyye Sarışahin, Researcher, Principal Investigator — Bezmialem Vakif University; Beyzanur Demirci, Researcher, Principal Investigator — Bezmialem Vakif University
Locations (1):
- Bezmialem Vakıf University, Istanbul, İ̇stanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
It will be shared with researchers who offer suggestions to improve the the study being carried out
Supporting Information: Study Protocol
Time Frame: 9 months
Access Criteria: Principal investigator will provide access.